CLINICAL TRIAL: NCT02095938
Title: Association of the Amisulpride Treatment Response in Patients With Schizophrenia With the Findings of Brain Structural Magnetic Resonance Imaging
Brief Title: Association of Amisulpride Response in Schizophrenia With Brain Image
Acronym: ARB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: CHA University (Other)
Collaborators: Handok Inc. (Industry)
Responsible Party: Principal Investigator, Sang-Hyuk Lee, Associate Professor, CHA University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Sang-Hyuk Lee; AMISUL06995 (Other Grant/Funding Number: Handok Inc.)
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia; Schizophreniform Disorder
Keywords: schizophrenia; brain structure; treatment response; solian; gene; mri
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Solian (Experimental): Amisulpride (Solian) will be orally administered once or twice daily after meal intake for 8 weeks. Patients initially will receive a low dose of amisulpride (200-400mg/day). The dosage may be adjusted to between 400 and 800mg/day according to the clinical decision by treating physician
  Interventions: Drug: amisulpride

INTERVENTIONS:
Drug: amisulpride — Amisulpride (Solian) will be orally administered once or twice daily after meal intake for 8 weeks. Patients initially will receive a low dose of amisulpride (200-400mg/day). The dosage may be adjusted to between 400 and 800mg/day according to the clinical decision by treating physician.
  Other Names: Solian

SUMMARY:
1. Study rationale - Nielsen et al reported that after 6 weeks of amisulpride treatment, patients with schizophrenia showed an increase in the anticipation-related functional MRI signal. This suggested that amisulpride could affect the brain structures and that responses to amisulpride could be associated by the brain structures as seen previous studies about treatment response to antipsychotics and brain structures. But to date, no study has examined the impact of brain structure alterations on amisulpride treatment for schizophrenia and its potential clinical significance.
2. Study Objectives 2-1. Primary: To show the differences of the baseline brain structures on the structural MRI between the Solian® treatment responders and the non-responders 2-2. Secondary: To show the differences of the baseline polymorphisms of COMT and BDNF with molecular genetic analysis between the Solian® treatment responders and the non-responders responder defined by PANSS. To find out the correlates of baseline brain structures with symptom severity of schizophrenia at baseline; symptom severity defined by CGI-S and PANSS. To assess psychotic symptom improvement after 8th week of Solian® treatment using PANSS, SANS, SAPS and CGI. To assess safety after 8th week of Solian® treatment with Barnes Akathisia Scale, Simpson-Angus scale and vital signs. To report all serious adverse event within 24hrs regardless of relationship to investigational product.
3. Study Design: Prospective/ Open label/ Interventional/ Controlled
4. Evaluation Criteria:

5-1. Primary endpoints: Brain structures on the structural MRI will be observed before the treatment starts. Based on the clinical response after treatment, patients will be divided in the two different groups as follow and their baseline brain structure of will be compared. Treatment responders and non-responders.

5-2. Secondary endpoints: The relationship of baseline brain structures with symptom severity of schizophrenia. Severity will be determined by CGI-S and PANSS at baseline. The differences of the polymorphisms of COMT and BDNF with molecular genetic analysis using patients' peripheral blood, especially leukocytes, between the treatment responders and the non-responders. Efficacy - PANSS, SANS, SAPS, CGI. Safety - Barnes akathisia scale, Simpson-Angus scale, Vital signs

DETAILED DESCRIPTION:
1. Study rationale 1-1.

   * Predicting the treatment response of antipsychotic drug in schizophrenia patients has been an issue in psychiatry. However, it is not clear if the findings of structural magnetic resonance imaging (MRI) such as brain gray matter volumes and white matter connectivities, are related to the treatment response of antipsychotic drugs.
   * The cognitive and behavioural symptoms of patients with schizophrenia are hypothesized to involve a disruption of neuronal interactions resulting in dysfunctional cognitive integration (Friston et al., 1995, 1996). This hypothesis is supported by reports about a decrease in white matter anatomic connections (Mitelman et al. 2006; Skudlarski et al. 2010; Zalesky et al. 2011) and brain structure alterations, especially decrease in volumes of specific brain regions for patients with schizophrenia. Several studies of brain connectivity have shown that functional connectivity depends strongly on the underlying anatomic structure (Sporns O et al. 2004). At the anatomic level, the pathology of schizophrenia has been related to a wide range of anatomic abnormalities, including ventricular enlargement, associated with anomalous neurodevelopment or neurodegenerative alterations (Shenton ME et al 2001). And schizophrenia is likely to be the result of both general and specific localized changes in both grey and white matter (Knochel C et al. 2012; Konrad A et al. 2008). Savas HA et al. found that responders to risperidone had greater hippocampal volumes than patients who failed to respond to risperidone (Savas HA et al., 2002). Vicente M et al. found an inverse association between striatal size and the degree of clinical improvement, and a direct association between the degree of insular volume deficit and its improvement. The non-responders to risperidone or olanzapine showed a significant decrease in their left rectal gyrus as compared with the responder group. (Vicente M et al., 2010).
   * Nielsen et al reported that after 6 weeks of amisulpride treatment, patients with schizophrenia showed an increase in the anticipation-related functional MRI signal (Nielsen et al., 2012). This suggested that amisulpride could affect the brain structures and that responses to amisulpride could be associated by the brain structures as seen previous studies about treatment response to antipsychotics and brain structures. But to date, no study has examined the impact of brain structure alterations on amisulpride treatment for schizophrenia and its potential clinical significance..
2. Study type: Clinical Study Phase IV
3. Number of centers: a single center in Korea
4. Number of subjects: N= 20 patients
5. Study duration and dates (format date : dd/mmm/yyyy) 5-1. Protocol planned date: 01/Apr/2013 5-2. First patient In: 01/Nov/2013 5-3. Last patient In: 01/Oct/2015 5-4. Last patient Out: 01/Dec/2015 5-5. Estimated enrollment duration: 2 years 5-6. Estimated average treatment duration: 8 weeks 5-7. Database lock planned date: 15/Dec/2015 5-8. Estimated Report/Publication date: 31/Dec/2015
6. Indication: Schizophrenia
7. Study Objectives (Primary / Most Important Secondary):

   7-1. Primary: To show the differences of the baseline brain structures on the structural MRI between the Solian® treatment responders and the non-responders 7-2. Secondary:
   * To show the differences of the baseline polymorphisms of COMT and BDNF with molecular genetic analysis between the Solian® treatment responders and the non-responders; responder defined by PANSS
   * To find out the correlates of baseline brain structures with symptom severity of schizophrenia at baseline; symptom severity defined by CGI-S and PANSS
   * To assess psychotic symptom improvement after 8th week of Solian® treatment using positive and negative syndrome scale (PANSS), scale for the assessment of negative symptoms (SANS), scale for the assessment of positive symptoms (SAPS) and clinical global impression scale (CGI)
   * To assess safety after 8th week of Solian® treatment with Barnes Akathisia Scale, Simpson-Angus scale and vital signs
   * To report all serious adverse event (SAE) within 24hrs regardless of relationship to investigational product. SAE or expedited reports are completed including: death, Requiring/prolonging hospitalization, Congenital anomaly/Birth defect, Life-threatening, Persistent/significant disability/incapacity, A procedure result only if symptomatic, considered by the investigator as clinically significant or meaningful or leading to permanent investigational product discontinuation or requiring corrective treatment, A symptomatic overdose, A pregnancy, AESI (adverse event special interest with immediate notification) in AEs( serious or non-serious) that need to be monitored, documented, and managed in a pre-specified manner described in the protocol.
8. Inclusion Criteria:

   8-1. between 21 and 60 years of age 8-2. diagnosed with schizophrenia, based on the Structured Clinical Interview for DSM-IV(SCID) 8-3. first or second episode of schizophrenia patient 8-4. the presence of positive or negative symptoms or both, resulting in illness of at least mild severity (≥3 on the Clinical Global Impression (CGI) severity scale
9. Exclusion Criteria:

   9-1. evidence of organic mental disorder or mental retardation 9-2. severe drug or alcohol dependence that required inpatient treatment and/or detoxification 9-3. other conditions, such as a serious medical condition, a history of bipolar or schizoaffective disorder, suicidality, possibility of pregnancy, lactation, or inability/unwillingness to use contraception 9-4. contraindicated with Solian® by the product label
10. Study Design: Prospective/ Open label/ Interventional/ Controlled
11. Treatments:

    11-1. Study medication - Solian® and there is no comparator medication. 11-2. Amisulpride (Solian) will be orally administered once or twice daily after meal intake for 8 weeks. Patients initially will receive a low dose of amisulpride (200-400mg/day). The dosage may be adjusted to between 400 and 800mg/day according to the clinical decision by treating physician.

    11-3. For efficacy assessment, psychotic symptoms will be assessed on baseline and 8th week by psychiatrists with positive and negative syndrome scale (PANSS), scale for the assessment of negative symptoms (SANS), scale for the assessment of positive symptoms (SAPS) and clinical global impression scale (CGI).

    11-4. For safety assessment, Barnes Akathisia Scale, Simpson-Angus scale and vital signs will be assessed on 8th week of treatment.

    11-5. Treatment responders will be defined as patients whose PANSS score reduction by 30% or more and patients whose PANSS score decrease by less than 30% will be assigned to non-responder group.

    11-6. The investigators will evaluate the differences of gray matter volume and white matter connectivity between responders and non-responders to amisulpride with images from brain 3T magnetic resonance imaging (MRI) using voxel-based morphometry (VBM) and tract-based spatial statistics (TBSS) at baseline. To examine a possible association between a specific brain region and response to amisulpride, the investigators will use methods based on the definition of regions of interest (ROIs).

    11-7. The investigators will evaluate the polymorphisms of COMT and BDNF with molecular genetic analysis using patients' peripheral blood, especially leukocytes at baseline. One-way analysis of variance (ANOVA) will be used to assess variations in clinical symptoms and cognitive function according to COMT and BDNF polymorphisms.
12. Evaluation Criteria:

    12-1 Primary endpoints
    * Brain structures on the structural MRI will be observed before the treatment starts. Based on the clinical response after treatment, patients will be divided in the two different groups as follow and their baseline brain structure of will be compared:
    * Treatment responders and non-responders; Treatment response will be defined as patients whose PANSS score reduce by 30% or more and non-responder as patients whose PANSS score decrease by less than 30% at 8 weeks from baseline.

    12-2 Secondary endpoints
    * The relationship of baseline brain structures with symptom severity of schizophrenia; Severity will be determined by CGI-S and PANSS at baseline.
    * The differences of the polymorphisms of COMT and BDNF with molecular genetic analysis using patients' peripheral blood, especially leukocytes, between the treatment responders and the non-responders
    * Efficacy : PANSS, SANS, SAPS, CGI on baseline and 8th week
    * Safety : Barnes akathisia scale, Simpson-Angus scale, Vital signs at 8th week
13. Study Budget 13-1. Total Study Cost (euro): 13,848 euro (1 EUR = 1445 KRW) 13-2. Y (year of Study Outline approval): 5,539 EUR 13-3. Y+1: 5,539 EUR 13-4. Beyond Y+1: 2,770 EUR

ELIGIBILITY:
Inclusion Criteria:

* between 21 and 60 years of age
* diagnosed with schizophrenia, based on the Structured Clinical Interview for DSM-IV(SCID)
* first or second episode of schizophrenia patient
* the presence of positive or negative symptoms or both, resulting in illness of at least mild severity (≥3 on the Clinical Global Impression (CGI) severity scale

Exclusion Criteria:

* evidence of organic mental disorder or mental retardation
* severe drug or alcohol dependence that required inpatient treatment and/or detoxification
* other conditions, such as a serious medical condition, a history of bipolar or schizoaffective disorder, suicidality, possibility of pregnancy, lactation, or inability/unwillingness to use contraception
* contraindicated with Solian® by the product label

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Brain structural MRI | baseline
  To show the differences of the baseline brain structures on the structural MRI between the Solian® treatment responders and the non-responders

SECONDARY OUTCOMES:
gene | baseline
  To show the differences of the baseline polymorphisms of COMT and BDNF with molecular genetic analysis between the Solian® treatment responders and the non-responders; responder defined by PANSS

OTHER OUTCOMES:
positive and negative syndrome scale | baseline, 8 week after treatment
  To assess psychotic symptom improvement after 8th week of Solian® treatment using positive and negative syndrome scale (PANSS), scale for the assessment of negative symptoms (SANS), scale for the assessment of positive symptoms (SAPS) and clinical global impression scale (CGI)
scale for the assessment of negative symptoms | baseline, 8 week after treatment
  To assess psychotic symptom improvement after 8th week of Solian® treatment using positive and negative syndrome scale (PANSS), scale for the assessment of negative symptoms (SANS), scale for the assessment of positive symptoms (SAPS) and clinical global impression scale (CGI)
scale for the assessment of positive symptoms | baseline, 8 week after treatment
  To assess psychotic symptom improvement after 8th week of Solian® treatment using positive and negative syndrome scale (PANSS), scale for the assessment of negative symptoms (SANS), scale for the assessment of positive symptoms (SAPS) and clinical global impression scale (CGI)
clinical global impression scale | baseline, 8 week after treatment
  To assess psychotic symptom improvement after 8th week of Solian® treatment using positive and negative syndrome scale (PANSS), scale for the assessment of negative symptoms (SANS), scale for the assessment of positive symptoms (SAPS) and clinical global impression scale (CGI)
Barnes Akathisia Scale | baseline, 8 week after treatment
  To assess safety after 8th week of Solian® treatment with Barnes Akathisia Scale, Simpson-Angus scale and vital signs
Simpson-Angus scale and vital signs | baseline, 8 week after treatment
  To assess safety after 8th week of Solian® treatment with Barnes Akathisia Scale, Simpson-Angus scale and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hyuk Lee, MD., PhD., Principal Investigator — Associate Professor at Bundang CHA hospital

REFERENCES:
- [Background] Friston KJ. Theoretical neurobiology and schizophrenia. Br Med Bull. 1996 Jul;52(3):644-55. doi: 10.1093/oxfordjournals.bmb.a011573. PMID 8949263
- [Background] Friston KJ, Frith CD. Schizophrenia: a disconnection syndrome? Clin Neurosci. 1995;3(2):89-97. PMID 7583624
- [Background] Knochel C, O'Dwyer L, Alves G, Reinke B, Magerkurth J, Rotarska-Jagiela A, Prvulovic D, Hampel H, Linden DE, Oertel-Knochel V. Association between white matter fiber integrity and subclinical psychotic symptoms in schizophrenia patients and unaffected relatives. Schizophr Res. 2012 Sep;140(1-3):129-35. doi: 10.1016/j.schres.2012.06.001. Epub 2012 Jul 19. PMID 22817874
- [Background] Konrad A, Winterer G. Disturbed structural connectivity in schizophrenia primary factor in pathology or epiphenomenon? Schizophr Bull. 2008 Jan;34(1):72-92. doi: 10.1093/schbul/sbm034. Epub 2007 May 7. PMID 17485733
- [Background] Mitelman SA, Newmark RE, Torosjan Y, Chu KW, Brickman AM, Haznedar MM, Hazlett EA, Tang CY, Shihabuddin L, Buchsbaum MS. White matter fractional anisotropy and outcome in schizophrenia. Schizophr Res. 2006 Oct;87(1-3):138-59. doi: 10.1016/j.schres.2006.06.016. Epub 2006 Jul 18. PMID 16854563
- [Background] Savas HA, Unal B, Erbagci H, Inaloz S, Herken H, Canan S, Gumusburun E, Zoroglu SS. Hippocampal volume in schizophrenia and its relationship with risperidone treatment: a stereological study. Neuropsychobiology. 2002;46(2):61-6. doi: 10.1159/000065413. PMID 12378121
- [Background] Shenton ME, Dickey CC, Frumin M, McCarley RW. A review of MRI findings in schizophrenia. Schizophr Res. 2001 Apr 15;49(1-2):1-52. doi: 10.1016/s0920-9964(01)00163-3. PMID 11343862
- [Background] Skudlarski P, Jagannathan K, Anderson K, Stevens MC, Calhoun VD, Skudlarska BA, Pearlson G. Brain connectivity is not only lower but different in schizophrenia: a combined anatomical and functional approach. Biol Psychiatry. 2010 Jul 1;68(1):61-9. doi: 10.1016/j.biopsych.2010.03.035. Epub 2010 May 23. PMID 20497901
- [Background] Sporns O, Chialvo DR, Kaiser M, Hilgetag CC. Organization, development and function of complex brain networks. Trends Cogn Sci. 2004 Sep;8(9):418-25. doi: 10.1016/j.tics.2004.07.008. PMID 15350243
- [Background] Molina V, Martin C, Ballesteros A, de Herrera AG, Hernandez-Tamames JA. Optimized voxel brain morphometry: association between brain volumes and the response to atypical antipsychotics. Eur Arch Psychiatry Clin Neurosci. 2011 Sep;261(6):407-16. doi: 10.1007/s00406-010-0182-2. Epub 2010 Dec 30. PMID 21191610
- [Background] Zalesky A, Fornito A, Seal ML, Cocchi L, Westin CF, Bullmore ET, Egan GF, Pantelis C. Disrupted axonal fiber connectivity in schizophrenia. Biol Psychiatry. 2011 Jan 1;69(1):80-9. doi: 10.1016/j.biopsych.2010.08.022. Epub 2010 Oct 29. PMID 21035793